CLINICAL TRIAL: NCT04951804
Title: A Randomized Controlled Trial of Endoscopic Ultrasound Guided Celiac Plexus Neurolysis (EUS-CPN) With and Without Bupivacaine
Brief Title: EUS-CPN With and Without Bupivacaine
Acronym: EUS-NB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21.151
Record Dates: First submitted 2021-06-09; First posted 2021-07-07 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Celiac plexus neurolysis; Bupivacaine; Endoscopic ultrasound; With Bupivacaine; Without Bupivacaine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-CPN with bupivacaine (Active Comparator): Endoscopic ultrasound guided celiac plexus neurolysis with absolute alcohol 20 mL preceded by injection of 10 ml of bupivacaine 0.5%.
  Interventions: Procedure: EUS-CPN with bupivacaine
- EUS-CPN without bupivacaine (Experimental): Endoscopic ultrasound guided celiac plexus neurolysis with absolute alcohol 20 mL only.
  Interventions: Procedure: EUS-CPN without bupivacaine

INTERVENTIONS:
Procedure: EUS-CPN without bupivacaine — Under conscious sedation, an echoendoscope is advanced into the stomach, just distal to the gastro-esophageal junction. The region of the celiac plexus is identified around the takeoff of the celiac artery from the aorta. Then, under real-time ultrasound guidance, a 19g needle is used to inject a neurolytic agent such as absolute alcohol around the base of the celiac artery.
  Arms: EUS-CPN without bupivacaine
Procedure: EUS-CPN with bupivacaine — Under conscious sedation, an echoendoscope is advanced into the stomach, just distal to the gastro-esophageal junction. The region of the celiac plexus is identified around the takeoff of the celiac artery from the aorta. Then, under real-time ultrasound guidance, a 19g needle is used to firstly inject bupivacaine and secondly a neurolytic agent such as absolute alcohol around the base of the celiac artery.
  Arms: EUS-CPN with bupivacaine

SUMMARY:
Endoscopic ultrasound (EUS) allows EUS-guided trans gastric injection of absolute alcohol around the base of the celiac plexus (celiac plexus neurolysis (EUS-CPN)), to help alleviate pain associated with pancreatic cancer.

It is standard procedure to inject bupivacaine immediately before injecting absolute alcohol, to theoretically prevent pain that may occur during and after the procedure. However, there are no data showing whether bupivacaine injection has any real influence on intra-procedural, immediate post-procedural, or long-term pain control. The injection of bupivacaine before the alcohol may have no effect, a synergistic effect, or an antagonistic effect, by diluting the alcohol, and reducing its neurolytic capacity. Inadvertent intravascular injection of bupivacaine may also cause irreversible cardiac arrhythmias and death.

The investigators therefore propose a randomized clinical trial to determine whether the exclusion of bupivacaine during EUS-guided CPN improves outcomes, or not.

DETAILED DESCRIPTION:
Pancreatic malignancies are the second most frequent gastrointestinal malignancy in Canada. From cancer mortality statistics in 2014, there were 4,700 new cases of pancreatic malignancies second only to colorectal cancer, representing 2.4% of all cancers. Even with chemotherapy, the median survival for patients with pancreatic adenocarcinoma is 6 to 10 months. Few patients are diagnosed at a resectable stage (12%-20%) so many patients are candidates for palliation only.

In this context, one of the most important symptoms is pain because it often affects both quality of life and survival. 70 to 80 % of patients with pancreatic cancer have abdominal pain at the time of diagnosis. Adequate pain control is therefore an essential component of care in these patients. In the initial phase, the pain is visceral, but with disease progression, somatic pain may occur, especially due to the peri-pancreatic invasion of neural structures, such as the celiac plexus.

Standard analgesics such as acetaminophen are usually ineffective and the use and effectiveness of opioids is frequently limited by side effects such as nausea, constipation, somnolence, confusion or respiratory depression.

The celiac plexus is immediately adjacent to the gastric wall. Endoscopic ultrasound (EUS) allows EUS-guided trans gastric injection of neurolytic agents around the celiac plexus (celiac plexus neurolysis [CPN]). Under conscious sedation, the echoendoscope is advanced into the stomach, just distal to the gastro-esophageal junction. The region of the celiac plexus is identified around the takeoff of the celiac artery from the aorta. Then, under real-time ultrasound guidance, a 19g needle is used to inject a neurolytic agent such as absolute alcohol around the base of the celiac artery. The entire procedure takes approximately 5 minutes. Absolute alcohol causes the immediate destruction of the celiac plexus neurons, by precipitation of endoneural lipoproteins and mucoproteins.

The effectiveness of CPN, is well established. It is safe, produces significant pain reduction, significantly reduces narcotic requirements, and may even increase survival. The investigators were the first to publish a randomized, sham-controlled trial demonstrating the efficacy of EUS-CPN for pain due to pancreatic cancer, and authored the most recent published guidelines on the use of EUS-CPN.

Based on our experience in over 1000 neurolysis procedures, patients undergoing EUS-guided CPN may experience pain, acutely during alcohol injection, and sometimes post-procedure, for up to a few hours. (Unpublished observations) It is possible that the presence of pain during injection of alcohol indicates that the celiac plexus has been accurately targeted and may therefore portend better long-term pain control.

Currently, during the neurolysis procedure, it is standard procedure to inject bupivacaine immediately before injecting absolute alcohol, to theoretically prevent pain during and after the procedure.

The true value of bupivacaine during neurolysis has never been studied. There are no data showing whether bupivacaine injection has any real influence on intra-procedural, immediate post-procedural, or long-term pain control. The injection of bupivacaine before the alcohol may have no effect, a synergistic effect, or an antagonistic effect, by diluting the alcohol, and reducing its neurolytic capacity. Inadvertent intravascular injection of bupivacaine may also cause irreversible cardiac arrhythmias and death.

In other words, in the worst case scenario, the injection of bupivacaine may increase procedural risk, without any associated benefit in terms of pain reduction.

The EUS team at the CHUM stopped using bupivacaine during neurolysis approximately 2 years ago and has noticed no obvious difference in pain during the procedure or in the immediate post-procedure recovery period, no increase in complications, and a possible reduction in requests for repeat neurolysis - suggesting that neurolysis without bupivacaine may be more effective. (Unpublished observations)

The investigators therefore propose a randomized clinical trial to determine whether the exclusion of bupivacaine during EUS-guided CPN improves outcomes, or not.

ELIGIBILITY:
Inclusion Criteria:

1. Malignant-appearing pancreatic mass, or proven pancreatic cancer involving the pancreatic genu, body, or tail
2. Any level of abdominal or back pain considered to be potentially related to the mass:

   1. New onset pain (<3 months)
   2. Constant
   3. Centrally located
   4. With or without irradiation to the back
   5. No obvious other source of pain based on history and physical examination by the attending endosonographer
3. No possibility of surgical management
4. Signed, informed consent
5. Celiac axis accessible for bilateral neurolysis at EUS.

Exclusion Criteria:

1. Allergy to bupivacaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Likert pain scores | Day 0 and Day 30
  Pain scale used : 7-point Likert scale for pain (minimum value is 0, maximum value is 6; higher scores mean a worse outcome)

SECONDARY OUTCOMES:
Difference in pain scores at T0 vs all other follow-up time points | Days 0, 3, 7, 30, 60, 90, 120
  The 7-point Likert scale for pain (minimum value is 0, maximum value is 6; higher scores mean a worse outcome)
Time to discharge from the endoscopy unit | From time of arrival in the recovery room after the intervention to time of discharge from the recovery room. The estimated period of time over which the event is assessed is up to two hours
  Time spent in the recovery room following the procedure
Narcotic usage | Narcotic usage for the 3 day-period preceding Days 0, 60 and 120
  Change in cumulative narcotic usage between Day 0 and Day 60, and between Day 0 and Day 120
Adverse events | Days 0, 3, 7, 30, 60, 90, 120
  Rate of all intervention-specific adverse events (Using the American Society of Gastrointestinal Endoscopy classification)
Survival | Up to 18 months
  Number of days between the EUS-CPN intervention and death
Difference in Global Rating Scale of Change at T3 vs all other follow-up time points | Days 3, 7, 30, 60, 90, 120
  The Global Rating Scale of Change will be used to measure subjects' impression of improvement in their health condition after T0 (the day celiac plexus neurolysis is performed) (minimum value is 0, maximum value is 6; higher scores mean a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: ANAND V SAHAI, MD, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal
Locations (1):
- Centre de recherche du Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Esmail E, Paquin SC, Sahai AV. Protocol for a randomized controlled trial of endoscopic ultrasound guided celiac plexus neurolysis (EUS-CPN) with vs without bupivacaine. Trials. 2023 Sep 8;24(1):576. doi: 10.1186/s13063-023-07487-7. PMID 37684697